CLINICAL TRIAL: NCT01348165
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 137882 in Healthy Male Volunteers (A Randomised, Single-blind, Placebo-controlled Phase I Study)
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 137882 in Healthy Male Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1306.1; 2010-023462-52 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-08

CONDITIONS: Healthy

ARMS (10):
- BI 137882 Dose 1 (Experimental): Powder for oral solution
  Interventions: Drug: BI 137882
- BI 137882 Dose 2 (Experimental): Powder for oral solution
  Interventions: Drug: BI 137882
- BI 137882 Dose 3 (Experimental): Powder for oral solution
  Interventions: Drug: BI 137882
- BI 137882 Dose 4 (Experimental): Powder for oral solution
  Interventions: Drug: BI 137882
- BI 137882 Dose 5 (Experimental): Powder for oral solution
  Interventions: Drug: BI 137882
- BI 137882 Dose 6 (Experimental): Powder for oral solution
  Interventions: Drug: BI 137882
- BI 137882 Dose 7 (Experimental): Powder for oral solution
  Interventions: Drug: BI 137882
- BI 137882 Dose 8 (Experimental): Powder for oral solution
  Interventions: Drug: BI 137882
- BI 137882 Dose 9 (Experimental): Powder for oral solution
  Interventions: Drug: BI 137882
- Placebo (Placebo Comparator): Powder for oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 137882 — Powder for oral solution
  Arms: BI 137882 Dose 1; BI 137882 Dose 2; BI 137882 Dose 3; BI 137882 Dose 4; BI 137882 Dose 5; BI 137882 Dose 6; BI 137882 Dose 7; BI 137882 Dose 8; BI 137882 Dose 9
Drug: Placebo — Powder for oral solution
  Arms: Placebo

SUMMARY:
Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 137882 in Healthy Male Volunteers

DETAILED DESCRIPTION:
As a transition from preclinical investigations to clinical development in this first-in-man trial, safety, tolerability, and pharmacokinetics of BI 137882 will be assessed in healthy male volunteers using single rising oral doses in order to provide the basis for a potential ongoing clinical development of BI 137882 in the indication of COPD.

Healthy male subjects aged 21 - 50 years will be recruited for this study. They provide a relatively stable physiological, biochemical and hormonal basis (steady state) for studying drug effects, they show no disease-related variation and they are not taking concomitant medication.

Within each dose group, all actively treated individuals will receive the same BI 137882 dose. The next higher dose will only be administered if the treatment in the preceding dose group was safe and well tolerated.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age 21 to 50 years
3. BMI 18.5 to 29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Smoker (more than 10 cigarettes /day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 20 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site
20. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms);
21. A history of additional risk factors for Torsades de points (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: A solution of 0.7% sodium dodecyl sulphate (SDS) and volume depends on corresponding dose group
- 0.01 mg: BI 137882 with 0.01 mg Dose level
- 0.03 mg: BI 137882 with 0.03 mg Dose level
- 0.1 mg: BI 137882 with 0.1 mg Dose level
- 0.25 mg: BI 137882 with 0.25 mg Dose level
- 0.5 mg: BI 137882 with 0.5 mg Dose level
- 0.6 mg: BI 137882 with 0.6 mg Dose level
Period: Overall Study
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Started | 10 | 5 | 6 | 6 | 6 | 1 | 6
Completed | 10 | 5 | 6 | 6 | 6 | 1 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set which included all subjects who received one dose of trial medication
Groups:
- Placebo: A solution of 0.7% SDS and volume depends on corresponding dose group
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg | Total
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 1 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (7.6) | 34.8 (10.3) | 40.8 (6.6) | 37.2 (7.1) | 36.5 (10.0) | 42.0 (NA) — Measure of variation not applicable as only one patient in treatment group | 35.5 (8.5) | 36.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 5 | 6 | 6 | 6 | 1 | 6 | 40
Smoking Status [Number; unit: participants]
  Never Smoked | 2 | 2 | 5 | 5 | 3 | 1 | 4 | 22
  Ex-Smoker | 3 | 2 | 1 | 0 | 2 | 0 | 0 | 8
  Currently Smokes | 5 | 1 | 0 | 1 | 1 | 0 | 2 | 10
Alcohol Status [Number; unit: participants] — Level of interference was based on if a subject drank alcohol to an extent that would interfere with the objectives of the trial.
  participants
    Never Drinker | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
    Drinks - no interference | 9 | 5 | 6 | 6 | 6 | 1 | 5 | 38
    Drinks - possible interference | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug Related Adverse Events
Description: Number of subjects with drug related adverse events (AEs)
Time Frame: From baseline up to 28 days
Population: Treated Set which included all subjects who received one dose of trial medication
Measure: Number; unit: Participants
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 1 | 6
Participants | 6 | 1 | 5 | 4 | 5 | 1 | 1

2. Primary Outcome: Blood Pressure
Description: Change from baseline for systolic blood pressure (SBP) and diastolic blood pressure (DBP)
Time Frame: Baseline and 28 days
Population: Treated Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 1 | 5
mmHg
  SBP | 1.0 (9.4) | 1.0 (3.4) | 2.8 (4.3) | -3.3 (6.9) | -5.8 (9.6) | -16 (NA) — Measure of dispersion not applicable as only one patient in this treatment group | 1.4 (7.0)
  DBP | -1.1 (3.7) | -1.6 (6.8) | -1.2 (2.7) | -2.2 (4.2) | -3.0 (3.7) | -12.0 (NA) — Measure of dispersion not applicable as only one patient in this treatment group | 0.8 (3.6)

3. Primary Outcome: Pulse Rate (PR)
Description: Change from Baseline to 28 Days in Pulse Rate
Time Frame: Baseline and 28 days
Population: Treated Set
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 1 | 5
bpm | 0.5 (12.8) | 6.4 (6.3) | 6.0 (5.8) | -0.7 (6.2) | 0.7 (5.2) | 3.0 (NA) — Measure of dispersion not applicable as only one patient in this treatment group | 0.8 (4.8)

4. Primary Outcome: Respiratory Rate (RR)
Description: Change from Baseline to 28 Days in Respiratory rate (RR)
Time Frame: Baseline and 28 days
Population: Treated Set
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 1 | 5
breaths/min | 0.3 (4.6) | 1.2 (5.4) | 1.3 (1.6) | 0.5 (2.1) | -1.8 (2.4) | 3.0 (NA) — Measure of dispersion not applicable as only one patient in this treatment group | 2.0 (3.2)

5. Secondary Outcome: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of BI 137882 in plasma.
Time Frame: 30 minutes (min) before drug administration and 30min, 1 hour (h), 2h, 4h, 6h, 8h, 12h, 24h, 34h, 48h, 72h, 96h, 144h, 192h, 264h, 336h and 480h after drug administration
Population: Treated Set. Descriptive statistics are only presented for treatment groups where the summary statistics were calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 6 | 6 | 6
nmol/L | 1.37 (20.0) | 4.79 (25.6) | 11.2 (21.7)

6. Secondary Outcome: Time to Maximum Measured Concentration (Tmax)
Description: Time from dosing to maximum measured concentration of the analyte in plasma.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 6 | 6 | 6
hours | 1.99 (68.8) [0.98 to 4.00] | 1.48 (62.9) [0.97 to 3.98] | 0.99 (115) [0.48 to 5.98]

7. Secondary Outcome: Area Under the Curve 0 to Infinity (AUC0-infinity)
Description: Area under the concentration-time curve of BI 137882 in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 6 | 6 | 6
nmol*h/L | 36.4 (19.6) | 153 (27.3) | 392 (25.2)

8. Secondary Outcome: Terminal Half-life (t1/2)
Description: Terminal half-life of BI 137882 in plasma.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 6 | 6 | 6
hours | 22.8 (17.7) | 35.8 (46.8) | 37.2 (27.0)

9. Secondary Outcome: Area Under the Curve 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 up to the last quantifiable data point.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 6 | 6 | 6
nmol*h/L | 14.6 (35.9) | 111 (27.5) | 348 (24.9)

10. Secondary Outcome: Terminal Rate Constant (λz)
Description: Terminal rate constant in plasma.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 6 | 6 | 6
1/h | 0.0304 (17.7) | 0.0194 (46.8) | 0.0186 (27.0)

11. Secondary Outcome: Mean Residence Time (MRTpo)
Description: Mean residence time of the analyte in the body after oral administration.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 6 | 6 | 6
hours | 32.9 (16.5) | 49.6 (41.1) | 52.8 (26.0)

12. Secondary Outcome: Apparent Clearance (CL/F)
Description: Apparent clearance of the analyte in plasma after extravascular administration.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 6 | 6 | 6
mL/min | 98.8 (19.6) | 58.7 (27.3) | 55.1 (25.2)

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Apparent volume of distribution of the analyte during the terminal phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 6 | 6 | 6
L | 195 (11.5) | 182 (28.2) | 177 (9.34)

14. Secondary Outcome: Amount of BI 137882 Eliminated in Urine From the Time Point t1 to Time Point t2
Description: Amount of BI 137882 eliminated in urine from the time point t1 to time point t2 (Aet1-t2)
Time Frame: 0-4, 4-8, 8-12, and 12-24 hours after drug administration
Population: There was no measurable BI 137882 excreted in urine so this pharmacokinetic parameter was not calculated.
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Fraction of BI 137882 Eliminated in Urine From Time Point t1 to Time Point t2
Description: Fraction of BI 137882 eliminated in urine from time point t1 to time point t2 (fet1-t2)
Time Frame: 0-4, 4-8, 8-12, and 12-24 hours after drug administration
Population: There was no measurable BI 137882 excreted in urine so this pharmacokinetic parameter was not calculated.
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Renal Clearance of BI 137882 From the Time Point t1 Until the Time Point t2
Description: Renal clearance of BI 137882 from the time point t1 until the time point t2 (CLR,t1-t2)
Time Frame: 0-4, 4-8, 8-12, and 12-24 hours after drug administration
Population: There was no measurable BI 137882 excreted in urine so this pharmacokinetic parameter was not calculated.
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Concentration of Tumour Necrosis Factor-alpha (TNF-α) Induced by Lipopolysaccharide (LPS) in Whole Blood ex Vivo
Description: Concentrations of TNF-α in plasma were determined by an enzyme-linked immunosorbent assay (ELISA). Concentrations of TNF-α in blood drawn after treatment with BI 137882 were compared with those in pre-dose samples to calculate the percent of inhibition of LPS induction of TNF-α production. Results indicate percent change from baseline of LPS-induced TNF-α production. A positive value indicates inhibition of the production.
Time Frame: 0.5 hours (h) before drug administration and 2h, 6h, 24h and 48h after drug administration
Population: Treated Set. Summary statistics were not calculated for the 0.5 mg group as there was only one patient in this group.
Measure: Mean (Standard Deviation); unit: percentage of TNF-α production
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
percentage of TNF-α production
  2 hours | -26.3 (45.0) | -23.1 (35.6) | -59.1 (35.9) | -23.9 (24.0) | 1.13 (20.0) | -0.41 (28.3)
  6 hours | 1.13 (64.5) | 37.9 (19.5) | -5.29 (34.7) | 11.4 (25.3) | -2.17 (60.5) | 12.8 (54.2)
  24 hours | -23.2 (41.8) | -11.6 (30.3) | 2.05 (20.7) | -16.4 (41.7) | 4.78 (36.5) | -17.1 (64.6)
  48 hours | -13.8 (44.3) | -3.90 (56.9) | 7.49 (33.0) | -61.0 (122) | -0.98 (22.6) | 3.52 (51.5)

18. Secondary Outcome: Concentration of Leukotriene B4 (LTB4) Induced by N-formyl-methionine-leucine-phenylalanine (fMLP) in Whole Blood ex Vivo.
Description: Percent of inhibition of fMLP induction of LTB4 production. Concentrations of LTB4 in plasma were determined by an enzyme-linked immunosorbent assay (ELISA). Results indicate percent change from baseline of fMLP induction of LTB4 production. A positive value indicates inhibition of the production.
Time Frame: 0.5 hours (h) before drug administration and 2h, 6h, 24h and 48h after drug administration
Population: Treated Set. Summary statistics were not calculated for the 0.5 mg group as there was only one patient in this group.
Measure: Mean (Standard Deviation); unit: percentage of LTB4 production
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
percentage of LTB4 production
  2 hours | -28.6 (47.3) | -0.83 (16.6) | 15.0 (29.8) | 11.1 (11.3) | -29.6 (35.6) | -74.4 (48.2)
  6 hours | 3.57 (44.7) | 5.26 (21.4) | 22.8 (29.5) | 5.92 (15.8) | -8.73 (39.3) | -69.1 (74.0)
  24 hours | -19.2 (58.1) | -19.1 (20.2) | -25.3 (27.8) | -12.1 (35.0) | -59.4 (66.4) | -61.2 (49.7)
  48 hours | -48.3 (89.7) | -38.1 (43.8) | -31.7 (23.2) | 1.11 (20.1) | -41.6 (54.3) | -94.2 (44.9)

19. Secondary Outcome: Area Under the Effect Curve (AUEC)
Description: Area under the effect curve for TNF-alpha induced by LPS and LTB4 induced by fMLP. Results indicate percent change from baseline of TNF-α/LTB4 production. A positive value indicates inhibition of the production.
Time Frame: 30 minutes (min) before drug administration and 2 hours (h), 6h, 24h and 48h after drug administration
Population: Treated Set. Summary statistics were not calculated for the 0.5 mg group as there was only one patient in this group. Geometric mean and geometric coefficient of variation was not calculated for any parameter in any dose group in which zero or a negative value was calculated, as geometric means cannot be calculated with negative or zero values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
pg*h/mL
  LPS | 25200 (85.9) | 34900 (221) | 10900 (654) | NA (NA) — No descriptive statistics calculated | 46900 (492) | 28700 (1050)
  fMLP | NA (NA) — No descriptive statistics calculated | NA (NA) — No descriptive statistics calculated | 25700 (6170) | 45100 (218) | NA (NA) — No descriptive statistics calculated | NA (NA) — No descriptive statistics calculated

20. Secondary Outcome: Maximum Effect (Emax)
Description: Maximum effect for TNF-alpha induced by LPS and LTB4 induced by fMLP. Results indicate percent change from baseline of TNF-α/LTB4 production. A positive value indicates inhibition of the production.
Time Frame: 30 minutes (min) before drug administration and 2 hours (h), 6h, 24h and 48h after drug administration
Population: Treated Set. Summary statistics were not calculated for the 0.5 mg group as there was only one patient in this group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
pg/mL
  TNF-alpha induced by LPS | 13400 (42.9) | 12000 (30.1) | 9990 (43.3) | 18200 (47.3) | 21500 (39.5) | 13800 (32.9)
  LTB4 induced by fMLP | 60400 (81.2) | 49400 (28.5) | 51300 (17.3) | 27800 (64.4) | 44800 (37.1) | 42100 (46.3)

21. Secondary Outcome: Minimum Effect (Emin)
Description: Minimum effect for TNF-alpha induced by LPS and LTB4 induced by fMLP. Results indicate percent change from baseline of TNF-α/LTB4 production. A positive value indicates inhibition of the production.
Time Frame: 30 minutes (min) before drug administration and 2 hours (h), 6h, 24h and 48h after drug administration
Population: Treated Set. Summary statistics were not calculated for the 0.5 mg group as there was only one patient in this group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 6
pg/mL
  TNF-alpha induced by LPS | 5200 (50.7) | 5500 (25.5) | 4730 (57.7) | 8210 (43.5) | 9570 (63.5) | 5890 (63.6)
  LTB4 induced by fMLP | 29000 (67.8) | 31100 (42.9) | 24000 (32.4) | 19000 (52.7) | 19500 (31.4) | 19900 (56.5)

22. Primary Outcome: Body Temperature
Description: Change from baseline to 28 Days in Body temperature
Time Frame: Baseline and 28 days
Population: Treated Set
Measure: Mean (Standard Deviation); unit: degrees celcius
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 1 | 5
degrees celcius | 0.0 (0.4) | 0.6 (0.4) | -0.3 (0.3) | 0.1 (0.5) | -0.3 (0.4) | -0.1 (NA) — Measure of dispersion not applicable as only one patient in this treatment group | 0.2 (0.5)

23. Primary Outcome: Assessment of Tolerability by Investigator
Description: The investigator assessed tolerability based on adverse events and the laboratory evaluation according to the categories 'good', 'satisfactory', 'not satisfactory', and 'bad'.
Time Frame: 28 days
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Number analyzed (Participants) | 10 | 5 | 6 | 6 | 6 | 1 | 5
Participants
  Good | 10 | 5 | 5 | 6 | 6 | 1 | 5
  Satisfactory | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Not satisfactory | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bad | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not assessable | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Until 5 days after drug administration
Description: Treatment emergent adverse events are presented, this excludes screening period and post treatment period.
Arm/Group | Placebo | 0.01 mg | 0.03 mg | 0.1 mg | 0.25 mg | 0.5 mg | 0.6 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/6 | 0/6 | 0/6 | 0/1 | 0/6
Other Adverse Events (participants affected / at risk) | 7/10 | 1/5 | 5/6 | 5/6 | 5/6 | 1/1 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | 0.01 mg (N=5) | 0.03 mg (N=6) | 0.1 mg (N=6) | 0.25 mg (N=6) | 0.5 mg (N=1) | 0.6 mg (N=6)
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypervigilance (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 3 | 2 | 2 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4 | 5 | 5 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The trial was put on hold due to a serious adverse event (post-treatment period) which was evaluated to be not drug related and the trial was subsequently terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes